CLINICAL TRIAL: NCT04278131
Title: Phase 1/2, Safety and Efficacy Trial of BS01, a Recombinant Adeno-Associated Virus Vector Expressing ChronosFP in Patients With Retinitis Pigmentosa
Brief Title: BS01 in Patients With Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionic Sight LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BS01-RP-001
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): BSO1 Cohort 1 dose
  Interventions: Drug: BS01
- Cohort 2 (Experimental): BS01 Cohort 2 dose
  Interventions: Drug: BS01
- Cohort 3 (Experimental): BS01 Cohort 3 dose
  Interventions: Drug: BS01
- Cohort 4 (Experimental): BS01 Cohort4 dose
  Interventions: Drug: BS01
- Cohort 5 (Experimental): BS01 Cohort4 dose
  Interventions: Drug: BS01
- Cohort 6 (Experimental): Treat opposite eye
  Interventions: Drug: BS01

INTERVENTIONS:
Drug: BS01 — Non-replicating, rep/cap-deleted, recombinant adeno-associated virus vector expressing an enhanced light-sensitive channelrhodopsin gene (ChronosFP)

SUMMARY:
A Phase 1/2, Safety and Efficacy Trial of BS01, a Recombinant Adeno-Associated Virus Vector Expressing ChronosFP (AAV2-CAG-ChronosFP) in Patients with Retinitis Pigmentosa

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of retinitis pigmentosa
* At least one eye with vision no better than 20/160 visual acuity on the EDTRS scale or, for patients with peripheral vision loss, a visual field no greater than 30°.

Exclusion Criteria:

* Prior receipt of any AAV gene therapy product
* Large amplitude nystagmus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 12 months
  Number of subjects with adverse events, changes in hematology/chemistry

SECONDARY OUTCOMES:
Secondary Outcome Measures | 12 months
  Changes in light detection (threshold to detect) Changes in motion detection Changes in shape/object/letter detection Changes in performance on maze navigation task

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Nirenberg, PhD, Study Director — Bionic Sight LLC
Locations (1):
- New Jersey Retina, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No